CLINICAL TRIAL: NCT06907355
Title: A Double-Blind Randomized Clinical Trial Comparing Levodropropizine, Codeine, Ivy Leaf (Hedera Helix Extract), and Placebo for the Treatment of Acute Cough in Adults With Upper Respiratory Tract Infections in Primary Care
Brief Title: CHAO Tos: Codeina, HederA Helix, LevOdropropizina Para la TOS
Acronym: CHAO TOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: UC CHRISTUS (Unknown)
Responsible Party: Principal Investigator, Diego Garcia Huidobro, Associate Professor, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 241001007
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Upper Resp Tract Infection
Keywords: Cough; Upper Respiratory Tract Infection; Levodropropizine; Codeine; Hedera Helix
MeSH Terms: conditions — Respiratory Tract Infections; Cough | interventions — Codeine; dipropizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Levodropropizine (Experimental): Levodropropizine 30mg/5ml: 10ml three times per day during 4 days
  Interventions: Drug: Levodropropizine
- Codeine (Experimental): Codeine 10mg/5ml + Pseudoephedrine 7.5mg/5ml + Chlorphenamine 0.5mg/5ml: 10ml three times per day during 4 days
  Interventions: Drug: Codeine
- Ivy Leaf (Hedera Helix Extract) (Experimental): Ivy Leaf (Hedera Helix Extract) 35 mg/5ml: 10ml three times per day during 4 days
  Interventions: Drug: Ivy Leaves Cough Liquid
- Placebo (Placebo Comparator): Vitamins: 10ml three times per day during 4 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Codeine — Codeine 10mg/5ml + Pseudoephedrine 7.5mg/5ml + Chlorphenamine 0.5mg/5ml: 10ml three times per day during 4 days
  Arms: Codeine
Drug: Levodropropizine — Levodropropizine 30mg/5ml: 10ml three times per day during 4 days
  Arms: Levodropropizine
Drug: Ivy Leaves Cough Liquid — Ivy Leaf (Hedera Helix Extract) 35 mg/5ml: 10ml three times per day during 4 days
  Arms: Ivy Leaf (Hedera Helix Extract)
Drug: Placebo — Vitamins: 10ml three times per day during 4 days
  Arms: Placebo

SUMMARY:
Upper respiratory tract infections affect millions globally, with cough being one of the most bothersome symptoms. While various treatments exist, their comparative effectiveness remains unclear. This study aims to evaluate and compare three commonly used treatments for acute cough in adults with upper respiratory tract infections: Levodropropizine, Codeine (with Pseudoephedrine and Chlorphenamine), and Ivy Leaf (Hedera Helix Extract). Investigators will conduct a double-blind, parallel-group randomized clinical trial with 184 adults aged 18-65 with acute upper respiratory tract infection and moderate to severe cough. Participants will be randomized to receive Levodropropizine, Codeine + Pseudoephedrine + Chlorphenamine, Ivy Leaf, or Placebo three times a day for 4 days. The primary outcome is cough severity at 48 hours, measured by a cough numerical rating scale. Secondary outcomes include cough severity and duration at 4- and 10-days. This trial will provide high-quality evidence comparing the efficacy of three widely used antitussive medications in primary care settings. The results could help establish evidence-based guidelines for treating acute cough in upper respiratory infections.

ELIGIBILITY:
Inclusion Criteria:

1. Have between 18 and 65 years of age.
2. Have an URTI with Jackson Score ≥6 points.
3. Have moderate or severe cough assessed by having a score ≥2 points in the cough domain of the Jackson Score and ≥60mm on the cough visual analogue scale (VAS).
4. Have initiated cough within 5 days of enrollment.
5. Be capable of understanding and complying with study procedures.
6. Sign a written informed consent.

Exclusion Criteria:

1. Physician considers that potential participant needs or might need to use antibiotics at the screening visit (e.g., suspected bacterial otitis, bacterial tonsilitis, bacterial sinusitis, bacterial bronchitis, or bacterial pneumonia) or suspected need for antibiotics during patient follow-up.
2. Individuals with pre-existing respiratory conditions, including asthma, chronic obstructive pulmonary disease (COPD), or any chronic lower respiratory tract disease.
3. Uncontrolled cardiovascular condition (hypertension, diabetes, etc.)
4. Contraindications to use Levodropropizine, Codeine, Pseudoephedrine, Chlorphenamine, or Ivy Leaf (Hedera Helix Extract), including Fructose Intolerance, Bronchorrhea, Kartagener Syndrome, Ciliary Dyskinesia, Respiratory Failure, Bronchial Obstructive Syndrome, severe Hypertension, Peptic Ulcer, using Monoamine Oxidase Inhibitors (MAOIs), CYP2D6 ultra-fast metabolizers.
5. Pregnancy, suspected pregnancy, desired pregnancy, or breastfeeding.
6. Contraindications to the study medications will also result in exclusion, including known or suspected allergies to Levodropropizine, Codeine, Pseudoephedrine, Chlorphenamine, or Hedera Helix Extract.
7. Known adverse reactions to Levodropropizine, Codeine, Pseudoephedrine, Chlorphenamine, or Hedera Helix Extract.
8. Participants currently using medications that could interfere with study outcomes, such as other cough suppressants, inhalers, or systemic corticosteroids.
9. Researcher considers participant might not comply with study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-11-22 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Change in cough severity | 48 hours
  Change in cough severity measured by a cough numerical rating scale (0-10, higher scores mean higher cough severity)

SECONDARY OUTCOMES:
Change in cough severity | 4 days
  Change in cough severity measured with the cough numerical rating scale (0-10, higher scores mean higher cough severity)
Change in cough severity | 10 days
  Change in cough severity measured with the cough numerical rating scale (0-10, higher scores mean higher cough severity)
Change in cough severity and duration | 48 hours
  Change in cough severity and duration measured with the Cough Severity Diary
Change in cough severity and duration | 4 days
  Change in cough severity and duration measured with the Cough Severity Diary
Change in cough severity and duration | 10 days
  Change in cough severity and duration measured with the Cough Severity Diary
Treatment failure | 4 days
  Categorical outcome:
  Yes: Persisting with a score ≥6 in the cough numerical rating scale (0-10) No: Not having cough or persisting with a score <6 in the cough numerical rating scale (0-10)
Treatment failure | 10 days
  Categorical outcome:
  Yes: Persisting with a score ≥6 in the cough numerical rating scale (0-10) No: Not having cough or persisting with a score <6 in the cough numerical rating scale (0-10)
Treatment safety | 48 hours
  Number of adverse events
Treatment safety | 4 days
  Number of adverse events
Treatment safety | 10 days
  Number of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Pontificia Universidad Catolica de Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided